CLINICAL TRIAL: NCT00277537
Title: A Phase III Multicenter, Randomised, Parallel, Placebo-Controlled, Double-Blind Study to Investigate the Safety and Efficacy of Treatment With Bronchitol (Dry Powder Mannitol) in the Symptomatic Treatment of Bronchiectasis.
Brief Title: Safety and Efficacy of Bronchitol in Bronchiectasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Syntara (Industry)
Responsible Party: Dr Brett Charlton, Pharmaxis Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DPM-B-301
Record Dates: First submitted 2006-01-13; First posted 2006-01-16 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-08

CONDITIONS: Bronchiectasis
Keywords: Mannitol
MeSH Terms: conditions — Bronchiectasis | interventions — Mannitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Mannitol
- 2 (Other)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Mannitol — 320mg BD 12 weeks followed by 40 weeks open label
  Arms: 1
Drug: placebo — BD for 12 weeks
  Arms: 2

SUMMARY:
Study will assess the safety and effectiveness of 12 week treatment with the study medication, Bronchitol, in subjects with bronchiectasis (a lung disease where patients have trapped, and often infected, thick, sticky mucus). Past studies have shown Bronchitol inhalation may help to facilitate the clearance of mucus by altering its rheology (making it less thick and sticky), thereby enhancing the shift of stagnant mucus from the lungs. On completion of the double blind phase, subjects will have the opportunity to participate in a 52 week open label phase.

ELIGIBILITY:
Inclusion Criteria:

* Non cystic fibrosis bronchiectasis
* Have FEV1 50% - 80% predicted and ≥1.0L
* Have chronic sputum production of >10 mL per day on the majority of days in the 3 months prior to study entry

Exclusion Criteria:

* Be using hypertonic saline or mucolytic pharmacological agents concurrently or in the 4 weeks prior to study entry
* Have airway hyperresponsiveness as defined by a positive Aridol challenge

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
24 hour sputum clearance | 24 hours / 12 weeks
Quality of Life SGRQ | 12 weeks

SECONDARY OUTCOMES:
bronchiectasis symptoms | 12 weeks
cough severity | 12 weeks
exercise capacity | 12 weeks
lung function, including gas transfer | 12 weeks
antibiotic use | 12 weeks
bronchial wall thickening and inflammation | 12 weeks
adverse events | 12 weeks / 12 months
haematology, biochemistry, | 12 weeks / 12 months
sputum microbiology quantitative and qualitative | 12 weeks / 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Brett Charlton, Study Director — Pharmaxis Ltd Australia
Locations (22):
- Australia (15):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown Sydney, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Bankstown Hospital, Sydney, New South Wales
  - Mater Adult Hospital, Brisbane, Queensland
  - Cairns Base Hospital, Cairns, Queensland
  - Repatriation General Hospital, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Burnside War Memorial Hospital, Toorak Gardens, Adelaide, South Australia
  - Peninsula Health Frankston Hospital, Frankston, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - AARI Sir Charles Gairdner Hospital, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (2):
  - Greenlane Hospital, Auckland
  - Middlemore Hospital, Auckland
- United Kingdom (5):
  - Belfast City Hospital, Belfast, Northern Ireland
  - Papworth Hospital, Cambridge
  - Glenfield Hospital, Leicester
  - North West Lung Centre, Wythshawe Hospital, Manchester
  - Norfolk and Norwich University Hospital, Norwich

REFERENCES:
- [Derived] Bilton D, Daviskas E, Anderson SD, Kolbe J, King G, Stirling RG, Thompson BR, Milne D, Charlton B; B301 Investigators. Phase 3 randomized study of the efficacy and safety of inhaled dry powder mannitol for the symptomatic treatment of non-cystic fibrosis bronchiectasis. Chest. 2013 Jul;144(1):215-225. doi: 10.1378/chest.12-1763. PMID 23429964